CLINICAL TRIAL: NCT03864601
Title: A Phase 1, Open-label Study to Determine the Absorption, Metabolism, and Routes of Excretion, Following Oral Administration of (14C) Radiolabeled JNJ-56136379 in Healthy Male Subjects
Brief Title: A Study of (14C) Radiolabeled JNJ-56136379 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR108586; 56136379HPB1007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-03-05; First posted 2019-03-06 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 14C-JNJ-56136379 (Experimental): Participants will receive a single oral 25 milligram (mg) dose of 14C-JNJ-56136379 on Day 1 under fed conditions.
  Interventions: Drug: 14C-JNJ-56136379

INTERVENTIONS:
Drug: 14C-JNJ-56136379 — 14C-JNJ-56136379 25 mg dose formulated as a polyethylene glycol (PEG)-based oral solution containing 3,145 kilo Becquerel (kBq) of 14C labeled JNJ-56136379, with a maximal total radiation burden of 1,000 micro Sievert.

SUMMARY:
The purpose of this study is to investigate the absorption, the metabolic pathways, the route and rate of elimination, and total recovery of 14C-JNJ-56136379 and/or total drug derived radioactivity in healthy male adult participants after administration of a single oral dose of 14C-JNJ-56136379.

ELIGIBILITY:
Inclusion Criteria:

* During the study (from the day of study drug intake onwards) and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving study drug, a male participant: must agree: (a) to wear a condom when engaging in any activity that allows for passage of ejaculate to another person (male participant should also be advised of the benefit for a female partner to use a highly effective method of contraception as condom may break or leak); (b) not to donate sperm for the purpose of reproduction.

Contraceptive use should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies

* Must have a body mass index (BMI; weight [kg]/height^2 [m]^2) between 18.0 and 30.0 kilogram per meter square (kg/m^2) (inclusive), and body weight not less than 50 kilogram (kg) at screening
* Healthy on the basis of physical examination, medical history and surgical history, and vital signs performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Healthy on the basis of clinical laboratory tests performed at screening
* Must have a normal 12-lead electrocardiogram (ECG) at screening

Exclusion Criteria:

* Any evidence of heart block or bundle branch block at screening
* Human immunodeficiency virus 1 (HIV-1) or HIV-2 infection (confirmed by antibodies) at screening
* History of hepatitis A, B, C, or E infection, or current hepatitis A infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]), or hepatitis B virus (HBV) infection (confirmed by hepatitis B surface antigen), or hepatitis C virus (HCV) infection (confirmed by HCV antibody), or hepatitis E infection (confirmed by hepatitis E [HEV] antibody IgM [in case HEV IgM positive, a confirmatory HEV ribonuclic acid {RNA} test should be performed]) at screening
* Any current, or history of, confirmed clinically significant skin disease requiring intermittent or chronic treatment such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, and urticaria
* A history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous studies with experimental drugs

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Cmax: Ratio of JNJ-56136379 Concentration and Total Radioactivity in Plasma | Up to 552 hours postdose
  Ratio of JNJ-56136379 concentration (plasma) and total radioactivity (plasma) for maximum observed plasma concentration (Cmax) will be assessed.
AUC(0-last): Ratio of JNJ-56136379 Concentration and Total Radioactivity in Plasma | Up to 552 hours postdose
  Ratio of JNJ-56136379 concentration (plasma) and total radioactivity (plasma) for area under the plasma concentration-time curve from time zero to last quantifiable concentration time (AUC[0-last]) will be assessed.
AUC(0-infinity): Ratio of JNJ-56136379 Concentration and Total Radioactivity in Plasma | Up to 552 hours postdose
  Ratio of JNJ-56136379 concentration (plasma) and total radioactivity (plasma) for area under the plasma concentration- time curve from time zero to infinite time (AUC [0-infinity]) will be assessed.
Total Radioactivity in Whole Blood, Plasma, Feces and Urine for 14C-JNJ-56136379 | Up to 552 hours postdose
  The total radioactivity of 14C-JNJ-56136379 in the whole blood plasma, feces and urine will be calculated.
Total Recovery of Radioactive Dose in Feces and Urine for 14C-JNJ-56136379 | Up to 552 hours postdose
  The amount of 14C-JNJ-56136379 recovered from the total administered radioactive dose in the feces and urine will be calculated.

SECONDARY OUTCOMES:
Metabolic Profiles of JNJ-56136379 in Plasma, Urine, and Feces | Predose (Day 1), 1, 2, 4, 8, 24, 48, 96, 192, 288, 432, 552 hours postdose (Day 24)
  The metabolite profiling of JNJ-56136379 in different matrices like plasma, urine, and feces will be performed and reported.
Maximum Observed Plasma Concentration (Cmax) of JNJ-56136379 | Predose (Day 1), 1, 2, 4, 8, 24, 48, 96, 192, 288, 432, 552 hours postdose (Day 24)
  Cmax is defined as the maximum observed plasma concentration.
Actual Sampling Time to Reach the Maximum Observed Plasma Concentration (Tmax) of JNJ-56136379 | Predose (Day 1), 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72, 96, 192, 288, 432, 552 hours postdose (Day 24)
  The Tmax is defined as actual sampling time to reach maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve from Time Zero to Last Quantifiable Concentration Time (AUC [0- Last]) of JNJ-56136379 | Predose (Day 1), 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72, 96, 192, 288, 432, 552 hours postdose (Day 24)
  AUC(0-Last) is area under the plasma concentration-time curve from time zero to time of the last measurable (non-below quantification limit) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration-Time Curve from Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-56136379 | Predose (Day 1), 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72, 96, 192, 288, 432, 552 hours postdose (Day 24)
  AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (last) and C(last)/lambda(z); where C(last) is the last observed measurable (non-below quantification limit) concentration.
Percentage of AUC(0-inifinity) (%AUC[0- infinity],ex of JNJ-56136379 | Predose (Day 1), 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72, 96, 192, 288, 432, 552 hours postdose (Day 24)
  %AUC(0-infinity).ex is the percentage of AUC obtained by extrapolation, calculated by the following equation: (AUC[0-inifinity] - AUC[0-last])/AUC(0-inifinity)*100.
Apparent Terminal Elimination Half-Life (t1/2) of JNJ-56136379 | Predose (Day 1), 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72, 96, 192, 288, 432, 552 hours postdose (Day 24)
  The t1/2 is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration time curve, and is calculated as 0.693/lambda(z).
Apparent Terminal Elimination Rate Constant (Lambda[z]) of JNJ-56136379 | Predose (Day 1), 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72, 96, 192, 288, 432, 552 hours postdose (Day 24)
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Amount of JNJ-56136379 Excreted in Urine within the Time Interval t1 to t2 (Ae[t1-t2]) | Predose and at every 24-hour interval up to 552 hours (Day 24) postdose
  Ae(t1-t2) is the amount of JNJ-56136379 excreted into urine for the collection interval from t1 to t2, where t1 and t2 are the start and end times of the interval, respectively, calculated by multiplying the urinary volume with the urinary concentration for that interval.
Amount of JNJ-56136379 Excreted in Urine (Ae) | Predose and at every 24-hour interval up to 552 hours (Day 24) postdose
  The Ae is the amount of JNJ-56136379 excreted in urine. It is calculated by multiplying the urinary volume with the urinary drug concentration.
Percentage of JNJ-56136379 Excreted in Urine (Ae%dose) | Predose and at every 24-hour interval up to 552 hours (Day 24) postdose
  The Ae%dose is the percentage of JNJ-56136379 dose excreted into the urine calculated as (Ae/dose)∗100.
Amount of JNJ-56136379 Excreted in Feces within the Time Interval t1 to t2 (Fe[t1-t2]) | Predose and at every 24-hour interval up to 552 hours (Day 24) postdose
  The Fe(t1-t2) is the amount of JNJ-56136379 excreted into feces for the collection interval from t1 to t2, where t1 and t2 are the start and end times of the interval, respectively, calculated by multiplying the fecal volume with the fecal concentration for that interval.
Amount of JNJ-56136379 Excreted in Feces (Fe) | Predose and at every 24-hour interval up to 552 hours (Day 24) postdose
  The Fe is the amount of JNJ-56136379 excreted in feces. It is calculated by multiplying the fecal volume with the fecal drug concentration.
Percentage of JNJ-56136379 Excreted in Feces (Fe,%dose) | Predose and at every 24-hour interval up to 552 hours (Day 24) postdose
  The Fe%dose is the percentage of JNJ-56136379 dose excreted into the feces calculated as (Fe/dose)*100.
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Approximately up to 2.5 months
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency